CLINICAL TRIAL: NCT05287061
Title: Implementation of a Positive Psychology Program in Cardiac Rehabilitation
Brief Title: Positive Psychology Program in Cardiac Rehabilitation
Acronym: PSICO-CARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Universitario 12 de Octubre (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17/171
Record Dates: First submitted 2022-03-11; First posted 2022-03-18 (Actual); Last update posted 2022-03-18 (Actual); Status verified 2022-03

CONDITIONS: Acute Coronary Syndrome
MeSH Terms: conditions — Acute Coronary Syndrome

STUDY DESIGN:
Intervention Model Description: Parallel group clinical trial, experimental group with psychological intervention versus control group without intervention
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cardiac Rehabilitation (CR) + Multicomponent Psychological Program (MPP): (Experimental): The patients who are assigned to this treatment arm will have access to a psychological intervention program, which will use techniques from the positive psychology and motivational interviewing to work on several modules: Health pills (phase I), CR in phase II identical to the standar, and MPP interspersed in Phase II of the conventional program. An individualized program will be included in this branch, which will be added to the follow-up carried out in primary care. It will contain a post-traumatic growth module, an emotion management module, and an intention consolidation module.
  Interventions: Behavioral: Multicomponent Psychological Program (MPP)
- Cardiac Rehabilitation (CR) (No Intervention): The patient will follow the usual process of cardiac rehabilitation.

INTERVENTIONS:
Behavioral: Multicomponent Psychological Program (MPP) — Patients will receive "health pills" during hospital admission. This intervention will be brief for individual application, but without specific content for each person, protocolized in its content and tools, and with a cognitive-behavioral orientation. Its therapeutic objective is to provide the patient with immediate control strategies for negative emotions and some pattern of active and positive coping. Two months after hospital discharge, the patients will also receive a multicomponent psychological program of a group nature. Based on motivational interviewing and positive psychology, with two blocks: emotions and consolidation of intentions. Two individual sessions will be carried out at the beginning to be able to do individual orientation, plan the intervention protocol, determine the objectives, the group intervention, and the specific action packages that the patient will receive.
  Arms: Cardiac Rehabilitation (CR) + Multicomponent Psychological Program (MPP):

SUMMARY:
Study to try to clarify the role of the dimensions of positive psychology as cardioprotective factors, controlling the classic CVR factors, both biomedical and psychosocial, as well as develop and test the effectiveness of a program Protocolized Psychological Intervention (PI), in a randomized clinical trial.

DETAILED DESCRIPTION:
It is intended to develop a collaborative study between Hospital Universitario 12 de October and the Faculty of Psychology of the Camilo José Cela University of Madrid to try to clarify the role of the dimensions of positive psychology as cardioprotective factors, controlling the classic CVR factors, both biomedical and psychosocial, as well as develop and test the effectiveness of a Protocolized Psychological Intervention, in a randomized clinical trial that will be developed in different phases of the cardiac recovery process in people who have had an acute coronary syndrome (ACS). The psychological intervention will include (1) a brief early intervention during hospitalization (based on psychoeducation, relaxation techniques, behavioral activation and focus on positive attitudes), and (2) during the follow-up phases, from two months after the hospital discharge, an intervention that will be made up of different packages depending on the individual profile (management of emotions, lifestyle healthy, post-traumatic growth and resilience, consolidation of intentions), versus a control group that will follow the standard cardiac rehabilitation program.

ELIGIBILITY:
Inclusion Criteria:

* Patients diagnosed with Acute Coronary Syndrome (ACS) referred to the CR Program and consent to participate in the trial.

Exclusion Criteria:

* Presence of diagnosed major psychiatric disorders according to DSM 5 criteria, who will be referred directly to the Psychiatry service.
* Inability to participate in a cardiac rehabilitation program for any reason.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 104 (Actual)
Dates: Start 2017-07-17 (Actual); Primary Completion 2018-07-01 (Actual); Study Completion 2019-07-01 (Actual)

PRIMARY OUTCOMES:
Level of Optimism | Week 10
  Measured by the Life Orientation Test - R (LOT-R; Scheier, Carver y Bridges, 1994
Level of Positive Emotions | Week 10
  Measured by the PERMA Questionnaire (Positive emotion, Engagement, Relationships, Meaning, and Accomplishment Questionaire; Seligman, 2011)
Level of Anxiety | Week 10
  Measured by the Hospital Anxiety and Depression Scale (Zigmond and Snaith, 1983)
Level of Depression | Week 10
  Measured by the Hospital Anxiety and Depression Scale (Zigmond and Snaith, 1983)
Level of Coping | Week 10
  Measured by the Brief-COPE Breve (Carver, 1997)
Level of Emotional Regulation | Week 10
  Measured by the Emotional Regulation Difficulties Scale (Gratz & Roemer, 2014)

CONTACTS AND LOCATIONS:
Overall Officials: Héctor Bueno, MD, PhD, Principal Investigator — Hospital Universitario 12 de Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Magan I, Jurado-Barba R, Moreno G, Ayan-Sanz MP, Izquierdo-Garcia J, Corradi G, Tello R, Bueno H. PsicoCare: a pilot randomized controlled trial testing a psychological intervention combining cognitive-behavioral treatment and positive psychology therapy in acute coronary syndrome patients. Front Psychol. 2024 Nov 19;15:1420137. doi: 10.3389/fpsyg.2024.1420137. eCollection 2024. PMID 39629185